CLINICAL TRIAL: NCT03629899
Title: Early Feasibility Study of the RETINA IMPLANT Alpha AMS in Blind Patients With Retinitis Pigmentosa
Brief Title: RETINA IMPLANT Alpha AMS in Blind Patients With Retinitis Pigmentosa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailability of the investigational device
Sponsor: Wills Eye (Other)
Collaborators: Retina Implant AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-645
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Inherited Retinal Degeneration; Retina Implant; Retinal Prosthesis; Artificial Vision
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- RETINA IMPLANT Alpha AMS (Experimental): After implantation surgery, every single sub-test will be performed with randomized implant activation ("ON" or "OFF"). During every trial of each sub-test there will be a study coordinator and a technician. The study coordinator will have a set randomization examination schedule while the technician will record patient response without knowledge of the randomization examination schedule. The patient, technician and investigator will all be masked to the testing conditions.
  Interventions: Device: RETINA IMPLANT Alpha AMS

INTERVENTIONS:
Device: RETINA IMPLANT Alpha AMS — Implantation of the subretinal RETINA IMPLANT Alpha AMS

SUMMARY:
The goal of this study is to transfer the surgical implantation technique and evaluate the safety and effectiveness of the RETINA IMPLANT Alpha AMS to restore limited visual function and functional vision in blind Retinitis Pigmentosa (RP) patients who are at the Light Perception (LP) or No Light Perception vision level (NLP). The safety of the implantation procedure and the long-term presence of the RETINA IMPLANT Alpha AMS will be assessed with clinical exams and objective clinical tests for the absence of any new permanent damage to the structure and function of the implanted eye with no permanent injury to the health and/or well being of the implanted patient as a result of the surgical procedure or presence of the implant. The effectiveness of the RETINA IMPLANT Alpha AMS will be evaluated by measuring limited visual function and functional vision in implanted subjects with the device "ON" and "OFF" in a randomized order. The ability to restore limited vision in blind RP patients with LP vision or NLP will reduce their disability and morbidity and provide a viable option to combat their disease and improve their lives.

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP) is a rare genetic disorder albeit the most common cause of inherited blindness. With progressive loss of function and cells in the outer retina, individuals with RP can progress to complete blindness of Light Perception or No Light Perception. There is no known cure or treatment for RP individuals at the Light Perception or No Light Perception phase of this progressive degenerative disease. The RETINA IMPLANT Alpha AMS is an investigational device designed to restore limited visual function and functional vision in this subset of patients suffering with RP whose visual acuity has deteriorated to the level of Light Perception or No Light Perception.

The RETINA IMPLANT Alpha AMS has been designed to replace the non-functioning and absent photoreceptor cells with a functional device to stimulate the remaining components of the retina to restore limited visual function and functional vision in patients with RP. The RETINA IMPLANT Alpha AMS device is surgically implanted subretinally to replace the non-functioning pathologic photoreceptor/RPE layer (or absent photoreceptor cells and defective pigment epithelium). The focusing lens system of the eye directs the visual image onto the device. When turned "ON" the device then stimulates the remaining visual cells of the inner layers of the retina and this visual information is subsequently transmitted by the remaining retinal network via the optic nerve to the visual cortex in the Central Nervous System (CNS).

This investigation is an Early Feasibility Study and will seek to implant five (5) to eight (8) patients. One surgical team, highly experienced in similar vitreoretinal procedures will be trained and will implant the enrolled patients. Follow-up visits for each patient will include an evaluation of safety and effectiveness at various time periods with follow-up continuing through five (5) years.

The use of masking in this clinical trial will be employed at the level of implanted subjects undergoing effectiveness evaluations during the follow-up visits as further described. Implant "ON" and "OFF" modality will be randomized and unknown to each subject undergoing functional vision tests during the follow-up visit. The "ON" and "OFF" will be encoded as either mode-1 or mode-2; for each test run, mode-1 and mode-2 will be differently encoded. The subject's visual performance will be evaluated and recorded for both "ON" and "OFF" implant conditions.

Each potential subject will undergo screening and evaluation to document that the eligibility criteria have been met and for proper surgical planning for implantation of the RETINA IMPLANT Alpha AMS. Qualifying subjects will undergo surgical implantation of the RETINA IMPLANT Alpha AMS in one eye and will be followed immediately in the post-operative period. Follow-up will continue for five (5) years.

ELIGIBILITY:
Inclusion Criteria:

• Blind RP patients with LP or NLP identified in both eyes using a photoflash test.

(NLP inclusion is defined as participants who at screening give less than 9 correct answers out of 20 trials to the photoflash test; LP inclusion is defined as participants who at screening give 9 or more correct answers out of 20 trials to the photoflash test)

* Pseudophakia for at least 3 months prior to entrance into study.
* Central visual function of 12 years / lifetime or greater with a history of reading vision in the eye to be implanted.
* Fluorescein angiography showing retinal vascular perfusion in all four quadrants of macula.
* Fifty (50) years of age or older at time of enrollment.
* Evidence of inner retinal function (ganglion cells and optic nerve function) by EEP test identified by the ability to elicit phosphene thresholds.
* ERG showing rod and cone non-function.
* Willing and able to give written informed consent and participate in ongoing follow-up.

Exclusion Criteria:

* Ophthalmic conditions other than RP with relevant effect upon visual function (e.g., glaucoma, optic neuropathies, trauma, diabetic retinopathy, retinal detachment, macular degeneration, cystoid macular edema, MS) with the addition of tobacco, alcohol abuse and retinotoxic drugs e.g. plaquenil and thorazine.
* Any other ocular disease that affects retina and / or optic nerve function.
* Opacification of ocular structures that prevent clear image transmission.
* Nystagmus.
* Cystoid macular edema within target region for implantation shown via Optical Coherence Tomography (OCT).
* Retina detected as too thin as shown via OCT (<100 μm) to expect required functionality of inner retina and /or OCT shows no layering of the inner retina in the central region.
* Scar tissue (e.g., epiretinal, intraretinal, subretinal, macular pucker) within target region for implantation.
* Heavily clumped pigmentation at posterior pole (would interfere with image transmission to vision chip).
* Anterior segment pathology that interferes with clear visualization of the retina (e.g., presence of cloudy or scarred cornea and / or papillary membrane) that cannot be resolved prior to entrance into study.
* Amblyopia reported earlier in life for eye to be implanted.
* Systemic diseases that might imply considerable risks with regard to the surgical interventions and anesthesia (e.g., cardiovascular / pulmonary diseases, severe metabolic diseases).
* Any condition and / or allergic contraindication to pre-operative, intra-operative, and post-operative medication.
* Health problems where general anesthesia is contraindicated.
* Disease or conditions that would probably limit life expectancy to less than 1 year from screening.
* Orbital deformity that would interfere with surgical implantation that could not be resolved prior to entrance into study.
* Patients with plastic intra-ocular lenses, or other materials, that would interact with silicone oil.
* Women who are pregnant or nursing, or women of childbearing potential who are not willing to use a medically acceptable means of birth control for the duration of the study, or women unwilling to perform a pregnancy test before entering the study.
* Neurological and / or psychiatric diseases (e.g., Parkinson, epilepsy, MS, depression or severe anxiety).
* Lack of cognitive and / or emotional ability (e.g., depression or severe anxiety) limiting participation as assessed by psychiatric evaluation.
* Participation in another interventional clinical trial within the past 30 days.
* The need for regular administration of anticoagulants, platelet aggregation inhibitors or analgesics containing acetylsalicylic acid.
* Disease or conditions that likely require regular use of MRI or other similar imaging technology that emits electromagnetic radiation.
* Patients unwilling to avoid participating in vigorous sports or activities with a high risk of a head injury.
* Patients unwilling to avoid security-scanning devices that would result in a full body, manual search.
* Ability to perceive form or motion under optimal conditions (largest size, brightest lighting, highest contrast, etc.) of form and motion testing as tested by BaLM, BaGA, and Landolt C.
* Patients with hearing deficits and cochlear implants or patients who may be implanted with cochlear implants in the near future.
* Patients undergoing or requiring medical treatments generating induced currents in the area of the implant such as electrosurgery, diathermy, neurostimulation, electroconvulsive therapy, ionizing radiation therapy, therapeutic ultrasound.
* Subjects with no active immunization status against organisms causing meningitis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of procedure or implant related adverse events | Through study completion, 5 years
  The safety endpoint is the absence of any new permanent damage to the function and structure of the implanted eye, consisting of new neovascularization, epiretinal membrane formation, and subretinal fibrotic tissue formation, and no permanent damage to the health and/or well-being of the subject following implantation as a result of the surgical procedure or presence of the implant.

SECONDARY OUTCOMES:
Change in visual function | Baseline, 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 52, 60 months post surgery
  Visual function will be assessed with the implant "ON" vs. "OFF" using Basic Light Localization and Motion Test (BaLM/BaGA).
Change in Visual Acuity | Baseline, 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 52, 60 months post surgery
  Change in visual acuity will be measured with the implant "ON" vs "OFF" using Landolt C-optotypes.
Changes in response to photoflash test | Baseline, 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 52, 60 months post surgery
  Changes in response to photoflash test
Change in Activities of Daily Living | Baseline, 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 52, 60 months post surgery
  Changes in daily life situations will be assessed in a real world environment with the implant "ON" vs "OFF"

CONTACTS AND LOCATIONS:
Overall Officials: Jay Federman, MD, Study Director — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stingl K, Schippert R, Bartz-Schmidt KU, Besch D, Cottriall CL, Edwards TL, Gekeler F, Greppmaier U, Kiel K, Koitschev A, Kuhlewein L, MacLaren RE, Ramsden JD, Roider J, Rothermel A, Sachs H, Schroder GS, Tode J, Troelenberg N, Zrenner E. Interim Results of a Multicenter Trial with the New Electronic Subretinal Implant Alpha AMS in 15 Patients Blind from Inherited Retinal Degenerations. Front Neurosci. 2017 Aug 23;11:445. doi: 10.3389/fnins.2017.00445. eCollection 2017. PMID 28878616
- [Background] Edwards TL, Cottriall CL, Xue K, Simunovic MP, Ramsden JD, Zrenner E, MacLaren RE. Assessment of the Electronic Retinal Implant Alpha AMS in Restoring Vision to Blind Patients with End-Stage Retinitis Pigmentosa. Ophthalmology. 2018 Mar;125(3):432-443. doi: 10.1016/j.ophtha.2017.09.019. Epub 2017 Oct 27. PMID 29110946